CLINICAL TRIAL: NCT07030309
Title: MEGA STUDY - Multicenter Evaluation of Gastroschisis Anomaly Study
Acronym: MEGA
Status: Active, not recruiting | Type: Observational
Sponsor: ResearchSkills (Network)
Responsible Party: Principal Investigator, Renata Jaczynska, Principal Investigator, ResearchSkills
Other Study IDs: 1/2025/MEGAStudy
Record Dates: First submitted 2025-05-03; First posted 2025-06-22 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Gastroschisis
Keywords: gastroschisis; ORPHA:2368; congenital anomaly; MEGA Study; Observational study; Epidemiology; Prenatal diagnosis; Multicenter study; prenatal ultrasound
MeSH Terms: conditions — Gastroschisis; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- simple gastroschisis: isolated gastroschisis, without intestinal anomalies
  Interventions: Other: Gastroschisis
- complex gastroschisis: gastroschisis with intestinal atresias, perforations, necrosis or volvulus
  Interventions: Other: Gastroschisis

INTERVENTIONS:
Other: Gastroschisis — Gastroschisis (GS) is a congenital abdominal wall defect in which the intestine is located outside the abdominal cavity. The prevalence of the GS classifies it as a rare disease (ORPHA:2368) Pregnancy complicated by gastroschisis is associated with an increased risk of serious perinatal complications.
  The presence of accompanying intestinal anomalies (atresia, necrosis, perforation, and volvulus), which qualifies the defect in the cGS (complex gastroschisis) group, as opposed to sGS (simple gastroschisis), where these anomalies are absent.
  cGS is associated with significantly increased neonatal morbidity and mortality when compared to sGS.

SUMMARY:
The purpose of this observational study is to evaluate selected epidemiological aspects of gastroschisis (GS) and factors affecting health outcomes of newborns with this diagnosis in a population of fetuses with gastroschisis. The main questions the study aims to answer are:

* Are there correlations between the parameters of ultrasound evaluation of the bowel with the condition of the newborn's bowel as assessed by the surgeon?
* What is the prevalence of the different forms of GS (classification according to the methodology of Molik et al. 2002, Perrone et al. 2018)?
* What is the incidence of perioperative and postoperative complications and other complications of the neonatal period?
* What is the relationship between the form of the defect (simple GS vs complex GS) and feeding milestones - TFEF, TPN, TSEF, TSOF, TFOF?
* What is the relationship between clinical parameters, diagnostic and therapeutic management, including method and timing of delivery, and final outcomes? Participants will not perform any active tasks or receive interventions as part of this study. Data will be collected passively from historical medical records including prenatal test results, details of pregnancy, delivery, and postnatal information on the newborn's treatment. The information collected will be anonymized. The study aims to collect information on prenatal diagnosis and neonatal outcomes, analyze factors affecting final results, and develop the most optimal management regimen for GS in Poland.

ELIGIBILITY:
Inclusion Criteria:

* A fetus with a diagnosis of gastroschisis;
* Availability of prenatal, delivery and postnatal records (for hospital discharge, transfer to another facility or death).

Exclusion Criteria:

* pregnancies terminated before the 22nd week of pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population for the MEGA Study consists of fetuses diagnosed with gastroschisis.
  The specific criteria for inclusion in the study are:
  * Fetuses with a diagnosis of gastroschisis.
  * Availability of prenatal, delivery, and postnatal documentation (up to hospital discharge, transfer to another center, or death).
  The exclusion criterion for the study is:
  • Pregnancies terminated before 22 weeks of gestation. The time frame for data included in the study is 2011 - 2024, although a shorter observation period may be applied depending on the availability of data at a participating center.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The prevalence of different forms of GS | During primary surgery
  The prevalence of different forms of GS: simple, complex

SECONDARY OUTCOMES:
Agreement rate between prenatal and neonatal assessment of the bowel condition | Prenatal assessment - during every US examination up to the time of delivery; newborn's evaluation - during primary surgery
  Comparison of the prenatal ultrasound bowel condition and the newborn's bowel assessment by the surgeon
Prevalence of necrotizing enterocolitis (NEC) | Up to 28 days after birth
  Diagnosis of necrotizing enterocolitis (NEC) is based on sudden onset of feeding intolerance, abdominal distention, bloody stools, and signs of sepsis (i.e., changes in the heart rate, respiratory rate, temperature, and blood pressure) in preterm infants, according to the Bell scale, which integrates the clinical and radiological manifestations.
Prevalence of short bowel syndrome (SBS) | During primary surgery or reoperation
  Diagnosis of short bowel syndrome (SBS) is in case of loss of bowel length or function significantly enough to cause malabsorption, requiring lifelong parenteral support
Prevalence of newborn sepsis | Up to 28 days after birth
  Newborn sepsis - an infection involving the bloodstream in infants under 28 days old. The clinical syndrome with symptomatology and laboratory findings consistent with a systemic inflammatory response to a multimodal infection caused by bacteria viruses, fungi potentially leading to multiple organ dysfunction, failure and even death within the first 28 days of life.
Time to full enteral feeding (TFEF) | From date of birth until the first day when full enteral feeding is achieved, assessed up to 28 days after birth.
  Time to full enteral feeding (TFEF) - the time when neonates start to receive all of their prescribed nutrition as milk feeds
Duration of the total parenteral nutrition (TPN) | From the first day of TPN initiation until the last day of TPN administration, assessed up to 28 days after birth.
  Total Parenteral Nutrition (TPN) - duration of parenteral nutrition, the time of intravenous feeding of nutritional products
Time to start enteral feeding (TSEF) | From date of birth until the first day enteral feeding is initiated, assessed up to 14 days after birth.
  Time to start enteral feeding (TSEF) - the time when neonates start enteral nutrition
Time to start oral feeding (TSOF) | From date of birth until the first day of oral feeding initiation, assessed up to 28 days after birth.
  Time to start oral feeding (TSOF)- the time when neonates start oral feeding
Time to full oral feeding (TFOF) | From date of birth until the first day full oral feeding is achieved, assessed up to 28 days after birth.
  Time to full oral feeding (TFOF) - the time to achieve oral exclusive feeding, without using additional or alternative feeding methods (such as gavage or nasogastric tube)
Lenght of hospital stay (LOS) | Time from the newborn's birth to discharge from the hospital, up to 28 days after birth
  Lenght of hospital stay (LOS) - duration of hospitalization - a clinical metric that measures the time elapsed between a patient's hospital admittance and discharge. For newborns - the time between the day of birth and its discharge
Prevalence of modes of delivery | At delivery
  Mode of delivery - method of pregnancy termination: vaginal delivery or cesarean delivery
Duration of pregnancy | At delivery
  Duration of pregnancy [days]
Time to repair (primary surgery) | From date and time of birth until the start of the primary surgical repair, up to 28 days after birth
  Time to repair (primary surgery); even primary closure or SILO [hours]
Time to closure abdominal wall defect | From date and time of birth until the completion of definitive abdominal wall defect closure, up to 28 days after birth
  Time to abdominal wall defect closure, even primary or secondary [hour]
Prevalence of neonatal death | Up to 28 days after birth
  Neonatal death within the first 28 days of life
Prevalence of intrauterine death | After 22 gestational weeks
  Intrauterine death after 22 gestational weeks
Prevalence of gastroschis types by Perrone et al. 2018 | During primary surgery, up to 28 days after birth
  Type A: ischemic bowel, significantly constricted at the ring without atresia Type B: ischemic bowel, significantly constricted at the ring (but viable) with an associated atresia Type C: ischemic bowel with a closing ring with nonviable external bowel (necrosis) with or without an associated atresia Type D: a completely closed defect with either a nubbin of exposed tissue or no external bowel
GPS (gastroschisis prognostic score) score by Cowan et al. 2012 | During primary surgery, up to 28 days after birth
  GPS (gastroschisis prognostic score) based on bowel appearance in newborns (within 6 hours of birth)
  I. Bowel matting:
  0 -none (normal bowel without inflammation)
  1. mild (slight inflammation or with a visible plaque on the surface (mild bowel matting), always needs to expand (required widening) the abdominal wall defect during primary closure)
  2. severe (moderate to massive inflammation with fibrous plaque (severe bowel matting) on the surface, stiffness of the intestinal wall EABL)
  II. Bowel atresia 0 - absent
  1. - suspected
  2. - present
  III. Bowel necrosis 0 - none
  1. focal
  2. - diffuse
  IV. Bowel perforation 0 - none 2 - present
Prevalence of Adverse Ultrasound Signs (AUS) | During every prenatal ultrasound examination, up to the time of delivery
  US 0-no adverse ultrasound signs: normal, stable, and adequate for the gestational age look of EABL (extra-abdominal bowel loops): normal bowel wall (non-hyperechoic, without oedema or/and thickening), free-floating loops without dilatation; no IABL (intra abdominal bowel loops) dilatation; no gastric dilatation.
  US 1-any ultrasound-adverse signs or progression: hyperechoic bowel wall or/and oedema or/and thickening; EABL dilatation; lack of lumen of EABL (collapsed bowel), non-free-floating loops with/or without bowel dilatation; IABL dilatation; gastric dilatation.
Prevalence of Fetal Growth Restriction (FGR) | Assessed throughout pregnancy, up to the time of delivery
  Fetal Growth Restriction (FGR) - "For early FGR (< 32 weeks), three solitary parameters (abdominal circumference (AC) < 3(rd) centile, estimated fetal weight (EFW) < 3(rd) centile and absent end-diastolic flow in the umbilical artery (UA)) and four contributory parameters (AC or EFW < 10(th) centile combined with a pulsatility index (PI) > 95(th) centile in either the UA or uterine artery) were agreed upon. For late FGR (≥ 32 weeks), two solitary parameters (AC or EFW < 3(rd) centile) and four contributory parameters (EFW or AC < 10(th) centile, AC or EFW crossing centiles by > two quartiles on growth charts and cerebroplacental ratio < 5(th) centile or UA-PI > 95(th) centile) were defined." Gordijn SJ, Beune IM, Thilaganathan B, Papageorghiou A, Baschat AA, Baker PN, Silver RM, Wynia K, Ganzevoort W. Consensus definition of fetal growth restriction: a Delphi procedure. Ultrasound Obstet Gynecol. 2016 Sep;48(3):333-9. doi: 10.1002/uog.15884.
Prevalence of Composite Intestinal Complications (CIC) | Up to 28 days after birth
  Composite Intestinal Complications (CIC) - intestinal complication (atresia, necrosis, perforation, volvulus) resulting from the definition of complex gastroschisis and peri-/post-operative complications in both forms (sGS and cGS) of defect (post-closure reoperation, adhesion-related bowel obstruction, bowel resection, Ileostomy/colostomy, the requirement to improve bowel anastomosis
Prevalence of bowel matting | During primary surgery, up to 28 days after birth
  Bowel matting: slight inflammation or with a visible plaque on the surface (mild bowel matting), always needs to expand (required widening) the abdominal wall defect during primary closure or moderate to massive inflammation with fibrous plaque (severe bowel matting) on the surface, stiffness of the intestinal wall EABL

CONTACTS AND LOCATIONS:
Overall Officials: Renata Jaczyńska, PhD, Principal Investigator — Uniwersyteckie Centrum Kliniczne Warszawskiego Uniwersytetu Medycznego [University Clinical Center Medical University of Warsaw]
Locations (9):
- Poland (9):
  - Górnośląskie Centrum Zdrowia Dziecka, Szpital Uniwersytecki ŚUM, Klinika Chirurgii Dziecięcej i Urologii Dziecięcej, Katowice
  - Szpital Kliniczny Uniwersytetu Medycznego w Poznaniu, Oddział Ginekologiczno-Położniczy, Pododdział Rozrodczości i Medycyny Perinatalnej, Poznan
  - Szpital Kliniczny Uniwersytetu Medyczny w Poznaniu, Klinika Chirurgii Traumatologii i Urologii Dziecięcej, Poznan
  - Szpital Miejski w Rudzie Śląskiej, Katedra i Oddział Kliniczny Ginekologii i Położnictwa, Wydziału Nauk o Zdrowiu, Ruda Śląska
  - Kliniczny Szpital Wojewódzki nr 2 im. Świętej Jadwigi Królowej. Klinika Położnictwa Ginekologii i Perinatologii, Rzeszów
  - Szpital Wojewódzki Nr 2 im. Św. Jadwigi Królowej w Rzeszowie, Klinika Chirurgii Dziecięcej, Rzeszów
  - Uniwersyteckie Centrum Kliniczne WUM, Dziecięcy Szpital Kliniczny. Klinika Chirurgii i Urologii Dziecięcej i Pediatrii, Warsaw
  - Instytut Matki i Dziecka, Warsaw
  - Uniwersyteckie Centrum Kliniczne Warszawskiego Uniwersytetu Medycznego. Klinika Położnictwa, Perinatologii, Ginekologii i Rozrodczości, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be analyzed for the purposes of the study but will not be shared. Only aggregate results will be published.
  Reason for not sharing IPD:
  The study protocol does not include plans for IPD sharing. Due to ethical considerations and data protection policies, only anonymized, group-level data will be included in publications and reports.

REFERENCES:
- [Background] Dekonenko C, Fraser JD, Deans KJ, Fallat ME, Helmrath M, Kabre R, Leys CM, Burns RC, Corkumd K, Dillon PA, Downard C, Wright TN, Gadepalli SK, Grabowski JE, Hernandez E, Hirschl R, Johnson KN, Kohler JE, Landman MP, Landisch RM, Lawrence AE, Mak GZ, Minneci PC, Rymeski B, Sato TT, Slater BJ, St Peter SD. Outcomes in gastroschisis: expectations in the postnatal period for simple vs complex gastroschisis. J Perinatol. 2021 Jul;41(7):1755-1759. doi: 10.1038/s41372-021-01093-8. Epub 2021 May 25. PMID 34035447
- [Background] Emil S, Canvasser N, Chen T, Friedrich E, Su W. Contemporary 2-year outcomes of complex gastroschisis. J Pediatr Surg. 2012 Aug;47(8):1521-8. doi: 10.1016/j.jpedsurg.2011.12.023. PMID 22901911
- [Background] Molik KA, Gingalewski CA, West KW, Rescorla FJ, Scherer LR, Engum SA, Grosfeld JL. Gastroschisis: a plea for risk categorization. J Pediatr Surg. 2001 Jan;36(1):51-5. doi: 10.1053/jpsu.2001.20004. PMID 11150437
- [Background] Burjonrappa S, Snyder AN. Regional variation in gastroschisis: a nationwide database review of demographics and outcomes. Pediatr Surg Int. 2021 Jul;37(7):911-917. doi: 10.1007/s00383-021-04894-2. Epub 2021 Mar 31. PMID 33787981
- [Background] Lap CCMM, Pistorius LR, Mulder EJH, Aliasi M, Kramer WLM, Bilardo CM, Cohen-Overbeek TE, Pajkrt E, Tibboel D, Wijnen RMH, Visser GHA, Manten GTR; FLAMINGO Study Working Group. Ultrasound markers for prediction of complex gastroschisis and adverse outcome: longitudinal prospective nationwide cohort study. Ultrasound Obstet Gynecol. 2020 Jun;55(6):776-785. doi: 10.1002/uog.21888. PMID 31613023
- [Background] Ferreira RG, Mendonca CR, Goncalves Ramos LL, de Abreu Tacon FS, Naves do Amaral W, Ruano R. Gastroschisis: a systematic review of diagnosis, prognosis and treatment. J Matern Fetal Neonatal Med. 2022 Dec;35(25):6199-6212. doi: 10.1080/14767058.2021.1909563. Epub 2021 Apr 25. PMID 33899664
- [Background] Arnold MA, Chang DC, Nabaweesi R, Colombani PM, Bathurst MA, Mon KS, Hosmane S, Abdullah F. Risk stratification of 4344 patients with gastroschisis into simple and complex categories. J Pediatr Surg. 2007 Sep;42(9):1520-5. doi: 10.1016/j.jpedsurg.2007.04.032. PMID 17848242
- [Background] South AP, Stutey KM, Meinzen-Derr J. Metaanalysis of the prevalence of intrauterine fetal death in gastroschisis. Am J Obstet Gynecol. 2013 Aug;209(2):114.e1-13. doi: 10.1016/j.ajog.2013.04.032. Epub 2013 Apr 26. PMID 23628262
- [Background] Bergholz R, Boettcher M, Reinshagen K, Wenke K. Complex gastroschisis is a different entity to simple gastroschisis affecting morbidity and mortality-a systematic review and meta-analysis. J Pediatr Surg. 2014 Oct;49(10):1527-32. doi: 10.1016/j.jpedsurg.2014.08.001. Epub 2014 Sep 4. PMID 25280661
- [Background] D'Antonio F, Virgone C, Rizzo G, Khalil A, Baud D, Cohen-Overbeek TE, Kuleva M, Salomon LJ, Flacco ME, Manzoli L, Giuliani S. Prenatal Risk Factors and Outcomes in Gastroschisis: A Meta-Analysis. Pediatrics. 2015 Jul;136(1):e159-69. doi: 10.1542/peds.2015-0017. PMID 26122809
- [Background] Wilson RD, Johnson MP. Congenital abdominal wall defects: an update. Fetal Diagn Ther. 2004 Sep-Oct;19(5):385-98. doi: 10.1159/000078990. PMID 15305094
- [Background] Benjamin B, Wilson GN. Anomalies associated with gastroschisis and omphalocele: analysis of 2825 cases from the Texas Birth Defects Registry. J Pediatr Surg. 2014 Apr;49(4):514-9. doi: 10.1016/j.jpedsurg.2013.11.052. Epub 2013 Nov 18. PMID 24726103
- [Background] Syngelaki A, Hammami A, Bower S, Zidere V, Akolekar R, Nicolaides KH. Diagnosis of fetal non-chromosomal abnormalities on routine ultrasound examination at 11-13 weeks' gestation. Ultrasound Obstet Gynecol. 2019 Oct;54(4):468-476. doi: 10.1002/uog.20844. PMID 31408229
- [Background] Garne E, Loane M, Dolk H, De Vigan C, Scarano G, Tucker D, Stoll C, Gener B, Pierini A, Nelen V, Rosch C, Gillerot Y, Feijoo M, Tincheva R, Queisser-Luft A, Addor MC, Mosquera C, Gatt M, Barisic I. Prenatal diagnosis of severe structural congenital malformations in Europe. Ultrasound Obstet Gynecol. 2005 Jan;25(1):6-11. doi: 10.1002/uog.1784. PMID 15619321
- [Background] Jones AM, Isenburg J, Salemi JL, Arnold KE, Mai CT, Aggarwal D, Arias W, Carrino GE, Ferrell E, Folorunso O, Ibe B, Kirby RS, Krapfl HR, Marengo LK, Mosley BS, Nance AE, Romitti PA, Spadafino J, Stock J, Honein MA. Increasing Prevalence of Gastroschisis--14 States, 1995-2012. MMWR Morb Mortal Wkly Rep. 2016 Jan 22;65(2):23-6. doi: 10.15585/mmwr.mm6502a2. PMID 26796490
- [Background] Prefumo F, Izzi C. Fetal abdominal wall defects. Best Pract Res Clin Obstet Gynaecol. 2014 Apr;28(3):391-402. doi: 10.1016/j.bpobgyn.2013.10.003. Epub 2013 Dec 3. PMID 24342556
- [Background] Jaczynska R, Mikulska B, Nimer A, Mydlak D, Sawicka E, Maciejewski T. Prenatal ultrasound markers for prediction of complex gastroschisis-single-center retrospective cohort study. J Perinatol. 2024 Sep;44(9):1325-1334. doi: 10.1038/s41372-024-02009-y. Epub 2024 Jun 19. PMID 38898181
- [Background] Jaczynska R, Mydlak D, Mikulska B, Nimer A, Maciejewski T, Sawicka E. Perinatal Outcomes of Neonates with Complex and Simple Gastroschisis after Planned Preterm Delivery-A Single-Centre Retrospective Cohort Study. Diagnostics (Basel). 2023 Jun 30;13(13):2225. doi: 10.3390/diagnostics13132225. PMID 37443619
- [Background] Youssef F, Laberge JM, Puligandla P, Emil S; Canadian Pediatric Surgery Network (CAPSNet). Determinants of outcomes in patients with simple gastroschisis. J Pediatr Surg. 2017 May;52(5):710-714. doi: 10.1016/j.jpedsurg.2017.01.019. Epub 2017 Jan 28. PMID 28188037
- [Background] Cowan KN, Puligandla PS, Laberge JM, Skarsgard ED, Bouchard S, Yanchar N, Kim P, Lee S, McMillan D, von Dadelszen P; Canadian Pediatric Surgery Network. The gastroschisis prognostic score: reliable outcome prediction in gastroschisis. J Pediatr Surg. 2012 Jun;47(6):1111-7. doi: 10.1016/j.jpedsurg.2012.03.010. PMID 22703779
- [Background] Sawicka E, Wieprzowski L, Jaczynska R, Maciejewski T. [Influence of selected factors on the treatment and prognosis in newborns with gastroschisis on the basis of own experience]. Med Wieku Rozwoj. 2013 Jan-Mar;17(1):37-46. Polish. PMID 23749694
- [Background] Nasr A, Langer JC; Canadian Paediatric Surgery Network. Influence of location of delivery on outcome in neonates with gastroschisis. J Pediatr Surg. 2012 Nov;47(11):2022-5. doi: 10.1016/j.jpedsurg.2012.07.037. PMID 23163992
- [Background] Apfeld JC, Kastenberg ZJ, Sylvester KG, Lee HC. The Effect of Level of Care on Gastroschisis Outcomes. J Pediatr. 2017 Nov;190:79-84.e1. doi: 10.1016/j.jpeds.2017.07.008. PMID 29144275
- [Background] Savoie KB, Huang EY, Aziz SK, Blakely ML, Dassinger S, Dorale AR, Duggan EM, Harting MT, Markel TA, Moore-Olufemi SD, Shah SR, St Peter SD, Tsao K, Wyrick DL, Williams RF. Improving gastroschisis outcomes: does birth place matter? J Pediatr Surg. 2014 Dec;49(12):1771-5. doi: 10.1016/j.jpedsurg.2014.09.019. Epub 2014 Nov 8. PMID 25487481
- [Background] Serra A, Fitze G, Kamin G, Dinger J, Konig IR, Roesner D. Preliminary report on elective preterm delivery at 34 weeks and primary abdominal closure for the management of gastroschisis. Eur J Pediatr Surg. 2008 Feb;18(1):32-7. doi: 10.1055/s-2007-965744. PMID 18302067
- [Background] Langer JC, Longaker MT, Crombleholme TM, Bond SJ, Finkbeiner WE, Rudolph CA, Verrier ED, Harrison MR. Etiology of intestinal damage in gastroschisis. I: Effects of amniotic fluid exposure and bowel constriction in a fetal lamb model. J Pediatr Surg. 1989 Oct;24(10):992-7. doi: 10.1016/s0022-3468(89)80200-3. PMID 2530329
- See also: Related Info — https://eu-rd-platform.jrc.ec.europa.eu